CLINICAL TRIAL: NCT04701931
Title: Topcon Maestro2 OCT Angiography Software Evaluation Study
Brief Title: OCT Angiography Software Evaluation Study
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THS-TPCN-2020-003
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-01

CONDITIONS: Retina Condition Followed by Fluorescein Angiography Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects presenting with Normal Eyes: Subjects with no known ocular diseases will be imaged on the Maestro2 OCT, Zeiss Cirrus HD-OCT 5000, and TRC-50DX
  Interventions: Device: Maestro2 OCTA; Device: Cirrus HD-OCT 5000; Device: TRC-50DX
- Subjects with retinal pathology present in the eye: Subjects with no known ocular diseases will be imaged on the Maestro2 OCT, Zeiss Cirrus HD-OCT 5000, and TRC-50DX
  Interventions: Device: Maestro2 OCTA; Device: Cirrus HD-OCT 5000; Device: TRC-50DX

INTERVENTIONS:
Device: Maestro2 OCTA — The Maestro2 OCTA with SS-OCT Angio software is an OCT with a fundus camera used for diagnostic purposes
Device: Cirrus HD-OCT 5000 — The Zeiss Cirrus HD-OCT 5000 is an OCT used for diagnostic purposes
Device: TRC-50DX — The TRC-50DX retinal camera images the fundus used for diagnostic purposes

SUMMARY:
Comparisons for vascular structure visualization in the retina and choroid.

DETAILED DESCRIPTION:
Evaluate the clinical performance of the Maestro2 OCTA for the visualization of the vascular structures of the retina and choroid.

ELIGIBILITY:
Pathology Population Inclusion Criteria

1. 22 years of age or older on the date of informed consent
2. Able to understand the written informed consent and willing to participate by signing the informed consent
3. Current diagnosis of one or more of the following pathologies in the study eye in two subgroups:

   1. Vascular pathologies primarily visualized in Superficial and Deep en face OCTA slabs, including but not limited to Diabetic Retinopathy (DR), Branch Retinal Vein Occlusion (BRVO), Central Retinal Vein Occlusion (CRVO), Central Retinal Arterial Occlusion (CRAO), Macular Telangiectasia (MacTel), Sickle Cell Retinopathy (SCR)
   2. Vascular pathologies primarily visualized in Outer Retina and Choriocapillaris en face OCTA slabs, including but not limited to Neovascular Age-Related Macular Degeneration ("wet" AMD) and Polypoidal Choroidal Vasculopathy (PCV) Exclusion Criteria

1. Subjects previously enrolled in Maestro2 OCTA feasibility study 2. Subjects who are pregnant or lactating* 3. Unable to complete the required clinical examinations 4. Contraindication to pupil dilation 6. Known allergy or other contradictions to fluorescein and/or to indocyanine green or iodides

Normal Population Inclusion Criteria

1. 22 years of age or older on the date of informed consent
2. Able to understand the written informed consent and willing to participate by signing the informed consent
3. BCVA 20/40 or better in the study eye Exclusion Criteria

1. Subjects previously enrolled in Maestro2 OCTA feasibility study 2. Subjects who are pregnant or lactating* 3. Unable to complete the required clinical examinations 4. Clinically significant findings in the study eye in clinical examination 5. Contraindication to pupil dilation 7. Known allergy or contradictions to fluorescein and/or to indocyanine green or iodides

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population with normal eye or eyes with pathology
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
OCTA image quality | Day 1
  The OCTA image quality comparison between Maestro2 and Cirrus
Visibility of key anatomical vascular features | Day 1
  The OCTA visibility comparison between Maestro2 and Cirrus
Identification of key pathological vascular features | Day 1
  the agreement rate is calculated based on the match outcome is the same between OCTA and FA/ICGA

CONTACTS AND LOCATIONS:
Overall Officials: Mayra Tafreshi, Study Director — CPAD
Locations (2):
- United States (2):
  - Orange County Retina Medical Group, Santa Ana, California
  - Southeast Retina Center, Augusta, Georgia